CLINICAL TRIAL: NCT00301808
Title: Phase II Study of Concurrent Cisplatin/Pemetrexed and RT Followed by Docetaxel in Stage III NSCLC (Non Small Cell Lung Cancer)
Brief Title: Cisplatin, Pemetrexed Disodium, and Radiation Therapy Followed by Docetaxel in Treating Patients With Stage III Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Shirish M. Gadgeel, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000461591; P30CA022453 (NIH); WSU-D-2934 (Other: Barbara Ann Karmanos Cancer Institute); WSU-0507002542 (Other: Wayne State University - Human Investigation Committee)
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Results first posted 2014-05-13 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2014-07

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Docetaxel; Pemetrexed; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cisplatin, Docetaxel & Radiation Therapy (Experimental): Cisplatin 75 mg/m2 every 3 weeks on days 1, 22, and 43; Docetaxel 75 mg/m2 on day 1 of each cycle; Radiation therapy will begin within 24 hours of the first cycle of chemotherapy.
  Interventions: Drug: Cisplatin; Drug: Docetaxel; Drug: Pemetrexed disodium; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 75 mg/m2 every 3 weeks on days 1, 22, and 43
  Other Names: Platin; Cisplatinum
Drug: Docetaxel — Docetaxel 75 mg/m2 on day 1 of each cycle
  Other Names: Taxotere®
Drug: Pemetrexed disodium — Pemetrexed 500 mg/m2 every 3 weeks on days 1, 22, and 43
  Other Names: Alimta
Radiation: Radiation therapy — Radiation therapy will begin within 24 hours of the first cycle of chemotherapy.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin, pemetrexed disodium, and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving more than one chemotherapy drug (combination chemotherapy) together with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving cisplatin and pemetrexed disodium together with radiation therapy followed by docetaxel works in treating patients with stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess 1-year survival of stage III non-small cell lung cancer (NSCLC) patients treated with cisplatin, pemetrexed disodium, and concurrent thoracic radiotherapy followed by consolidation therapy with docetaxel.

Secondary

* Assess the progression-free survival and overall survival.
* Assess the toxicity of this regimen.

OUTLINE: Patients receive pemetrexed disodium IV over 10 minutes followed by cisplatin IV over 60 minute on day 1. Treatment repeats every 21 days for 3 courses in the absence of unacceptable toxicity. Patients also receive concurrent thoracic radiotherapy in weeks 1-7. Between 3-8 weeks after completion of chemoradiotherapy, patients with no progressive disease receive docetaxel IV over 1 hour on day 1. Treatment with docetaxel repeats every 21 days for 3 courses.

After completion of study therapy, patients are followed at 1 month and periodically thereafter.

PROJECTED ACCRUAL: A total of 28 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologic or cytologic diagnosis of non-small cell lung cancer (NSCLC), meeting 1 of the following staging criteria:

  * Stage IIIA disease, meeting all of the following criteria:

    * Mediastinal lymph node involvement

      * Greater than one mediastinal lymph node enlarged on CT scan, confirmed by positron emission tomography (PET) scan
    * Paralyzed left vocal cord with separate lung primary distinct from the aorto-pulmonary lymph nodes on the CT scan
  * Stage IIIB disease, meeting all of the following criteria:

    * N3 lymph node involvement

      * Enlarged N3 lymph nodes on CT scan confirmed by PET scan

        * Lymph node involvement may not extend to cervical lymph nodes other than supraclavicular lymph nodes
    * Right-sided primary tumor with left vocal cord paralysis
    * Evidence of tumor extension into the mediastinum and/or mediastinal structures by mediastinoscopy, bronchoscopy, or CT scan
    * No evidence of malignant pleural effusion unless effusion is only evident on CT scan
    * No more than 1 parenchymal lesions on the same or opposite sides of the lung
* No brain metastases by CT scan or MRI

PATIENT CHARACTERISTICS:

* SWOG performance status 0 or 1
* Platelet count ≥ 100,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Creatinine clearance ≥ 45 mL/min
* Bilirubin normal
* Transaminases (SGOT and/or SGPT) ≤ 1.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Total lung volume (i.e., right and left lung minus the gross tumor volume) receiving greater than 20 Gy of radiation ≤ 40%
* FEV_1 ≥ 70% of predicted
* DLCO ≥ 50 mL/min
* No other concurrent malignancy

  * Prior malignancy allowed provided it is in clinical control and is not likely to impact clinical outcome in the opinion of the treating physician
* No peripheral neuropathy ≥ grade 2
* No serious medical illness, including, but not limited to, any of the following:

  * Uncontrolled congestive heart failure
  * Uncontrolled angina
  * Myocardial infarction
  * Cerebrovascular event within the past 6 months
  * History of chronic active hepatitis
  * History of HIV infection
  * Active bacterial infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Must be willing and able to take folic acid, cyanocobalamin (vitamin B12), or dexamethasone

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy for NSCLC
* No concurrent participation in another therapeutic investigational study
* Concurrent ibuprofen (400 mg four times daily) allowed during pemetrexed disodium administration provided the patient has normal renal function
* No concurrent aspirin or other nonsteroidal antiinflammatory drugs (NSAIDs) 2 days before, during, and for 2 days after pemetrexed disodium administration

  * Patients on long-acting NSAIDs (e.g. naproxen sodium, diflunisal, nabumetone, or celecoxib) must be willing or able to discontinue usage 5 days prior to, during, and for 2 days after pemetrexed disodium administration

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2005-11; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shirish M. Gadgeel, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (2):
- United States (2):
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan

REFERENCES:
- [Derived] Gadgeel SM, Ruckdeschel JC, Patel BB, Wozniak A, Konski A, Valdivieso M, Hackstock D, Chen W, Belzer K, Burger AM, Marquette L, Turrisi A. Phase II study of pemetrexed and cisplatin, with chest radiotherapy followed by docetaxel in patients with stage III non-small cell lung cancer. J Thorac Oncol. 2011 May;6(5):927-33. doi: 10.1097/JTO.0b013e3182156109. PMID 21415776

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cisplatin, Docetaxel & Radiation Therapy
Started | 29
Completed | 17
Not Completed | 12
Not completed — Adverse Event | 5
Not completed — Death | 3
Not completed — Lack of Efficacy | 4

BASELINE CHARACTERISTICS:
Arm/Group | Cisplatin, Docetaxel & Radiation Therapy
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.76 (8.03)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Probability of Overall Survival at One Year
Description: Overall Survival at one year using Kaplan-Meier product-limit analysis
Time Frame: at 1 year
Measure: Number (95% Confidence Interval); unit: probability of overall survival at 1 yr.
Arm/Group | Cisplatin, Docetaxel & Radiation Therapy
Number analyzed (Participants) | 29
probability of overall survival at 1 yr. | 0.66 [0.48 to 0.84]
Statistical Analysis 1: Comparison: Cisplatin, Docetaxel & Radiation Therapy; Test type: Superiority or Other; Kaplan-Meier product limit = 0.66, 95% CI 2-sided [0.48 to 0.84], Standard Error of Mean .1423

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival using Kaplan-Meier estimates
Time Frame: Approximately 3 weeks after the last cycle of cisplatin/pemetrexed or completion of radiation whichever is the later.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cisplatin, Docetaxel & Radiation Therapy
Number analyzed (Participants) | 29
months | 16.9 [7.2 to 36.2]

3. Secondary Outcome: Overall Survival
Description: Overall survival using Kaplan-Meier estimates
Time Frame: Date of registration to the date of death
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cisplatin, Docetaxel & Radiation Therapy
Number analyzed (Participants) | 29
months | 33.7 [6.4 to NA] — All observations after the median was reached are censored.

4. Secondary Outcome: Safety Outcomes
Description: Toxicity: total number of SAEs and other AEs
Time Frame: 72 hours after 2nd and 3rd cycles: 30 days after completion of study treatment; Every 2 months thereafter; then once a year
Measure: Number; unit: Adverse event
Arm/Group | Cisplatin, Docetaxel & Radiation Therapy
Number analyzed (Participants) | 29
Adverse event
  Serious (grade 3 or 4) | 20
  other (grade 0, 1, or 2) | 245

ADVERSE EVENTS:
Time Frame: Approximately 7 years
Arm/Group | Cisplatin, Docetaxel & Radiation Therapy
Serious Adverse Events (participants affected / at risk) | 15/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cisplatin, Docetaxel & Radiation Therapy (N=29)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fever (General disorders) | 2 (2)
Acute renal failure (Renal and urinary disorders) | 3 (3)
Hypotension (Vascular disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Chronic obstructive pulmonary exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cisplatin, Docetaxel & Radiation Therapy (N=29)
Esophagitis (Gastrointestinal disorders) | 20 (20)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Decreased WBC count (Investigations) | 22 (22)
Anemia (Blood and lymphatic system disorders) | 22 (22)
Neutropenia (Blood and lymphatic system disorders) | 17 (17)
Platelet count decreased (Investigations) | 17 (17)
Fatigue (General disorders) | 20 (20)
Fever (General disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 13 (13)
Vomiting (Gastrointestinal disorders) | 11 (11)
Anorexia (Metabolism and nutrition disorders) | 14 (14)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 25 (25)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Alkaline phosphatase increased (Investigations) | 2 (2)
Alanine Aminotransferase (ALT) (Investigations) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 6 (6)
Creatinine increased (Investigations) | 6 (6)
Infection (Infections and infestations) | 6 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4)
Pain (General disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)

LIMITATIONS AND CAVEATS:
Study being a single institution, single arm study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No